CLINICAL TRIAL: NCT06840431
Title: Randomized Control Trial of the Co-Parenting for Resilience Program
Acronym: CPR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ronald Cox, Professor of Human Develop and Family Science, Oklahoma State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Oklahoma State University; 1R15HD112895-01 (NIH)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Child Wellbeing
Keywords: divorce; child wellbeing; co-parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In person condition (Experimental): This condition tests program effects when delivered by a trained non-clinical facilitator.
  Interventions: Behavioral: in-person condition
- online condition (Experimental): This condition tests program effects when the program is delivered asynchronously online
  Interventions: Behavioral: online condition
- Self-help book with quiz (Placebo Comparator): This condition serves as a placebo control comparing the intervention components to a knowledge only condition.
  Interventions: Behavioral: self-help condition

INTERVENTIONS:
Behavioral: in-person condition — participants will receive program components in a classroom setting with a trained non-clinical facilitator.
  Arms: In person condition
Behavioral: online condition — Participants will receive program components in an asynchronous online format.
  Arms: online condition
Behavioral: self-help condition — Participants will read a self-help book on how to manage their divorce and take a quiz to ensure that the book has been read.
  Arms: Self-help book with quiz

SUMMARY:
Because parental divorce has been linked to a significant increase in mental health diagnoses among children, it is important to develop effective interventions that reduce the negative impact of divorce on children. This study assesses the efficacy of the Co-Parenting for Resilience (CPR) resilience program by randomly assigning divorcing individuals to three different forms of the intervention to test whether one or both of versions of CPR are better than reading a self-help book, and whether an in-person version of CPR is more effective than an online version. The three conditions or versions are: 1) an in-person version of CPR taught by a trained non-clinician, 2) an asynchronous fully online version of CPR, and 3) a group that simply reads a self-help book and responds to a knowledge check to ensure the material was read.

DETAILED DESCRIPTION:
Reducing the effects of parental divorce on children is a clear but often overlooked public health issue. Nearly 44% of the 66 million children living in the U.S. will experience their parents' divorce or separation by age 15. Because children whose parents divorce are more likely to develop social, emotional, behavioral and physical problems and have lower academic performance than their peers from intact families; and because more children of divorce (25%) are diagnosed with mental illness compared to children in the general population (10%), addressing the negative impacts of divorce on children is a national imperative.

Parental management of the divorce process has been shown to be key in determining child adjustment, with greater mismanagement and conflict associated with multiple negative outcomes for children. Divorce can create considerable turmoil in people's lives leading some parents to mishandle their own emotions. Highly emotional parents often place their children in the middle of their conflict, overly rely on children to meet their own emotional needs, or practice avoidance coping through alcohol and drugs or by otherwise abandoning their children. Divorce education programs claiming to help parents ameliorate the effects of divorce on children abound in all 50 states; and over half of states mandate attendance by statute. However, recent reviews reveal major weaknesses in program development and evaluation, such as: (a) few programs are guided by theories of behavior change and only seek to increase knowledge; (b) the majority of programs have not been evaluated, and those that have lack methodological rigor; (c) child outcomes are rarely assessed either directly or indirectly through parent report, (d) important moderators to help determine for whom the program is effective (e.g., parent gender and ethnicity, low- vs. high-conflict couples, reasons for divorce) have not been explored; and (e) although online programs proliferated during COVID-19, they have largely not been tested. Addressing these and other weaknesses is critical to making scientific progress in the field and to developing programs with demonstrated efficacy in helping the millions of parents and children avoid the more severe effects of divorce.

The Co-Parenting for Resilience (CPR) program innovatively merges research from Family Therapy and Prevention Science to address many of the above-mentioned weaknesses. CPR is a 4-hour psychoeducational intervention that draws from empirically supported approaches such as Brief Strategic Family Therapy, Motivational Interviewing, and Family Stress Theory, and uses a combination of instruction, interactive activities, and guided reflections to promote the deep learning and paradigm shifts that aid in changing maladaptive cognitions and in promoting effective parenting and improved child outcomes. Initial findings from a pilot study suggest that CPR reduces parent reports of conflict and stress and increases parental collaboration, hope, and parent reports of child adjustment. These findings, however, were based on a quasi-experimental design with a non-equivalent control group. The proposed R15 project advances the science by leveraging a long-standing partnership with the Oklahoma County District Court to conduct a 3-arm RCT that will accomplish three specific aims:

1. Determine the relative efficacy of the online and in-person versions of CPR to improve child post-divorce adjustment compared to each other and to a bibliotherapy control group at 3- and 12-month follow-ups.
2. Test paths from the online and in-person versions of CPR to child adjustment via parenting competencies.
3. Identify moderators of the effectiveness of in-person and online formats of CPR such as parent gender, ethnicity, and level and type of conflict between divorcing partners.

Primary hypotheses tested are that the effects of CPR on child post-divorce adjustment will: (H1) be higher in both CPR conditions relative to the control group; (H2) not differ between the two CPR conditions; (H3) be mediated by parenting competencies, and (H4) there will be moderation by level and type of conflict.

We will randomly assign 300 unique individuals (not couples) who have filed for divorce to one of the three arms (n=100 each arm). Data will be collected at three timepoints: baseline (pre-intervention), at 3-months to test for program efficacy and mediation, and at a 12-month follow-up controlling for baseline. Participants will be parents of either gender who are filing for divorce with a child from 4-10 years old.

Per the R15 mechanism, this project proposes three objectives: (1) to conduct a small-scale research project whose aims address a significant public health issue, the physical and mental health of divorcing parents and their children; (2) to expose graduate and undergraduate students to different phases of the research process; and (3) to expand institutional research capacity.

The project will innovatively: 1) leverage the court system to rigorously answer questions significant to science and to divorcing families, 2) test an online version of the CPR program that will benefit an underserved rural population, 3) inform further program development by identifying key program moderators, and 4) provide critical empirical evidence for the dissemination of the CPR program to other states.

ELIGIBILITY:
Inclusion Criteria:

* One adult member of a dyad filing for a divorce or legal separation (e.g., non-married couples) in Oklahoma County with a biological minor child aged 4-10,
* Being an English or Spanish speaker,
* Having internet access necessary for the online group (necessary for this randomized trial.
* In the event participants have more than one child, they will be asked to report on their oldest child with the person they are divorcing who is age 10 or under. Focus on the oldest child counterbalances the age distribution of children expected per our preliminary data, thereby facilitating a test of age differences in treatment effects.

Exclusion Criteria:

* Parents under the age of 18,
* Parents who do not consent to randomization,
* Parents who are illiterate.
* Only one member of the dyad will be allowed in the study.
* We also exclude parents for whom the target child is not the biological child of both parents. Stepfamilies, adoptive families, grandparents raising grandchildren, and other family types have dynamics not directly comparable to families with two biological parents and is beyond the scope of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | Baseline, 3-month follow-up, and 12-month follow-up
  The SDQ is a widely used measure consisting of 25 items that make up five subscales on which parents report their child's emotional symptoms, conduct problems, hyperactivity, peer problems, and prosocial behavior. The SDQ has been normed on children from 4-17 years of age and provides a total child difficulty score and a score for each of the five subscales. For our primary analyses of child adjustment, we will use the total child difficulty score.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Cox, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Sharing individualized data rather than aggregate data would be a breach of confidentiality and is not permitted by our IRB.

REFERENCES:
- [Background] Cox, R.B., et al., Hope, Stress, and Post-Divorce Child Adjustment: Development and Evaluation of the Co-Parenting for Resilience Program. Journal of Divorce & Remarriage, 2021. 62(2): p. 144-163.
- [Background] Hill, R., Generic features of families under stress. Social Casework, 1958. 39(2-3): p. 139-150.
- [Background] Hill, R., Families under stress: Adjustment to the crises of war separation and return. 1949.
- [Background] Miller, W.R. and S. Rollnick, Motivational interviewing: Helping people change. 2012: Guilford press.
- [Background] Fisch, R., J. Weakland, and L. Segal, The tactics of change: Doing therapy briefly. 1982, San Francisco: Jossey-Bass.
- [Background] Sigal A, Sandler I, Wolchik S, Braver S. Do Parent Education Programs Promote Healthy Post-Divorce Parenting? Critical Distinctions and a Review of the Evidence. Fam Court Rev. 2011 Jan;49(1):120-139. doi: 10.1111/j.1744-1617.2010.01357.x. PMID 21552360
- [Background] Kierstead, S., Parent education programs in family courts: Balancing autonomy and state intervention. Family Court Review, 2011. 49(1): p. 140-154.
- [Background] Pollet, S.L. and M. Lombreglia, A nationwide survey of mandatory parent education. Family Court Review, 2008. 46(2): p. 375-394.
- [Background] Dunn J, Davies LC, O'Connor TG, Sturgess W. Family lives and friendships: the perspectives of children in step-, single-parent, and nonstep families. J Fam Psychol. 2001 Jun;15(2):272-87. PMID 11458633
- [Background] Sandler I, Gunn H, Mazza G, Tein JY, Wolchik S, Berkel C, Jones S, Porter M. Effects of a Program to Promote High Quality Parenting by Divorced and Separated Fathers. Prev Sci. 2018 May;19(4):538-548. doi: 10.1007/s11121-017-0841-x. PMID 28913663
- [Background] Amato, P.R., The consequences of divorce for adults and children: An update. Drustvena istrazivanja, 2014. 23(1): p. 5-24.
- [Background] Andersson, G., E. Thomson, and A. Duntava, Life-table representations of family dynamics in the 21st century. Demographic Research, 2017. 37: p. 1081-1230.
- [Background] Vezzetti VC. New approaches to divorce with children: A problem of public health. Health Psychol Open. 2016 Nov 15;3(2):2055102916678105. doi: 10.1177/2055102916678105. eCollection 2016 Jul. PMID 28070408